CLINICAL TRIAL: NCT01456143
Title: In Vivo Multimodal Imaging of Upper Aerodigestive Epithelia
Brief Title: Optical Imaging of Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left, study to be re-open with new PI, no planned data analysis
Sponsor: Sharmila Anandasabapathy, MD (Individual)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor-Investigator, Sharmila Anandasabapathy, MD, Principal Investigator, Anandasabapathy, Sharmila, M.D.
Organization: Anandasabapathy, Sharmila, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 09-2057
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Squamous Cell Carcinoma; Neoplasia; Head and Neck Cancer
Keywords: Squamous Cell Carcinoma; Neoplasia; Optical imaging; Head and Neck Cancer; Oropharynx; Larynx; Oral Cavity
MeSH Terms: conditions — Carcinoma, Squamous Cell; Neoplasms; Head and Neck Neoplasms; Laryngeal Diseases | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HRME with proflavine (Experimental): High Resolution Microendoscopy (HRME) imaging device that operates as a fluorescence microscope with a fiber optic imaging probe. The probe is placed against the mucosa to obtain images relayed to a tablet computer. 0.01% Proflavine hemisulfate used as a fluorescent contrast agent applied topically to mucosa. HRME is used to capture images of suspicious areas sprayed with proflavine hemisulfate.
  Interventions: Device: High Resolution Microendoscopy (HRME); Other: Proflavine hemisulfate

INTERVENTIONS:
Device: High Resolution Microendoscopy (HRME) — High Resolution Microendoscopy imaging device that operates as a fluorescence microscope with a fiber optic imaging probe. The probe is placed against the mucosa to obtain images relayed to a tablet computer.
  Other Names: HRME
Other: Proflavine hemisulfate — 0.01% Proflavine hemisulfate used as a fluorescent contrast agent applied topically to mucosa
  Other Names: Proflavine

SUMMARY:
This study examines if certain imaging techniques and devices can aid the surgeon in detecting cancer during the surgical procedure.

DETAILED DESCRIPTION:
The purpose of this study is to determine if optical imaging modalities used at the time of surgical resection for head and neck squamous cell carcinoma can help delineate normal from cancerous mucosa. The High resolution microendoscope, developed by our collaborators at Rice university, can allow for real time visualization of tissue nuclei. The overall aim of this study is to determine if this device can be used to enhance the accuracy of intraoperative margin detection during tumor resection for head and neck cancer.

At the time of tumor resection for head and neck squamous cell carcinoma, a wide field imaging device will be used to identify suspicious areas. The High resolution device will then image representative areas from the tumor, the tumor margin, and normal mucosa. A topical dye, proflavin, will be placed on the tissue to enhance the visualization of nuclei prior to imaging with the HRME device. Following imaging, biopsies of the imaged areas will be taken and submitted for pathology diagnosis. The images of the biopsies will then be compared and the device will be evaluated for accuracy of margin detection at the time of tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy Proven Squamous Cell Carcinoma of the oral cavity, oropharynx, larynx, hypopharynx
* Must be receiving surgical treatment for their cancer

Exclusion Criteria:

* Presence of medical or psychiatric condition affecting the ability to give informed consent
* Known allergy to Proflavin
* Pregnant or nursing Females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sikora, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sharmila Anandasabapathy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HRME With Proflavine
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HRME With Proflavine Hemisulfate: High Resolution Microendoscopy imaging device used in conjunction with proflavine hemisulfate as a contrast agent
Arm/Group | HRME With Proflavine Hemisulfate
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.09 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Accuracy
Description: Accuracy of reviewers in differentiating neoplastic or benign mucosa in comparison to the pathology results
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Mean (95% Confidence Interval); unit: Percent of images with correct diagnosis
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
Percent of images with correct diagnosis | 95.1 [94 to 96]

2. Primary Outcome: Sensitivity
Description: Sensitivity = probability that the HRME correctly classifies as positive those with neoplasia compared to pathology results
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Mean (95% Confidence Interval); unit: Percent of images with correct diagnosis
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
Percent of images with correct diagnosis | 96 [94 to 99]

3. Primary Outcome: Specificity
Description: Specificity = Probability that the HRME correctly classifies as negative those without neoplasia compared to pathology results
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Mean (95% Confidence Interval); unit: Percent of images with correct diagnosis
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
Percent of images with correct diagnosis | 95 [90 to 99]

4. Primary Outcome: Positive Predictive Value
Description: PPV = proportion of those with a positive test who have neoplasia compared to pathology results
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Mean (95% Confidence Interval); unit: Percent of images with correct diagnosis
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
Percent of images with correct diagnosis | 91 [85 to 98]

5. Primary Outcome: Negative Predictive Value
Description: NPV = proportion of those with a negative test without neoplasia compared to pathology results
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Mean (95% Confidence Interval); unit: Percent of images with correct diagnosis
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
Percent of images with correct diagnosis | 98 [97 to 99]

6. Primary Outcome: Interrater Reliability
Description: Amount of agreement among the 11 blinded head and neck cancer specialists, determined by the Fleiss Kappa. 33 benign and 65 cancer images were evaluated by the reviewers who were blinded to the anatomical site, tumor subsite, and final histopathologic diagnosis. Each reviewer was asked to classify each image as benign or neoplastic. The reviewers evaluated the images based on nuclear size, nuclear to cytoplasmic ratio, and overall cell architecture. Images were randomized in their presentation to the reviewers as to not establish any pattern. Each reviewer provided their interpretation in isolated settings to avoid influence from other reviewers.
Time Frame: Immediately following image (day of enrollment or up to 2 weeks after enrollment)
Measure: Number (95% Confidence Interval); unit: proportion of agreement among 11 experts
Arm/Group | HRME With Proflavine
Number analyzed (Participants) | 33
proportion of agreement among 11 experts | .81 [.78 to .84]

ADVERSE EVENTS:
Time Frame: (day of enrollment or up to 2 weeks after enrollment)]
Description: Serious and other adverse events were monitored and assessed, but none were observed
Arm/Group | HRME With Proflavine Hemisulfate
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No